CLINICAL TRIAL: NCT04037540
Title: Comparison of Conservative and Operative Treatment of Jones Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-KUCH-01-Jones; CZ.02.1.01/00/00/17_049/00084 (Other Grant/Funding Number: Ministry of Education of the Czech Republic)
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Fracture of Fifth Metatarsal Bone
Keywords: Jones fracture; The American Orthopaedic Foot & Ankle Society (AOFAS); Herbert screw

STUDY DESIGN:
Intervention Model Description: The patients with Jones fracture were randomized into one of the two study groups - operational or conservative approach.
Masking Description: No masking was used in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Operational approach (Experimental): The patients enrolled in this arm underwent surgical treatment of the Jones fracture.
  Interventions: Procedure: Operational approach
- Conservative approach (Experimental): The patients enrolled in this arm were treated conservatively, using fixation of the injured extremity.
  Interventions: Procedure: Conservative approach

INTERVENTIONS:
Procedure: Operational approach — Operational approach was used to treat the Jones fracture in patients randomized into the respective study arm.
  Arms: Operational approach
Procedure: Conservative approach — Conservative approach was used to treat the Jones fracture in patients randomized into the respective study arm.
  Arms: Conservative approach

SUMMARY:
The study deals with the topic of treatment of Jones fracture, comparing surgical and conservative approach. The fracture occurs especially in highly active individuals.

DETAILED DESCRIPTION:
The study deals with the topic of treatment of Jones fracture, comparing surgical and conservative approach. The fracture occurs especially in highly active individuals.

The study proposes a supposition of recommending the active operational approach, which shortens the period of healing by 6 weeks, limitation of physical activity by 4 weeks, and sick leave by 2 months. It also completely eliminates the need to perform a rigid fixation of the extremity for 8-12 weeks.

ELIGIBILITY:
Inclusion Criteria:

- Jones fracture

Exclusion Criteria:

* combined injury
* recurring injury
* diabetes mellitus
* chronic renal insufficiency
* osteopathy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2011-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The American Orthopaedic Foot & Ankle Society (AOFAS) score - 6 weeks | 6 weeks
  The improvement in The American Orthopaedic Foot & Ankle Society (AOFAS) score from the baseline was observed at 6 weeks after injury on a scale of 0-100.
AOFAS score - 12 months | 12 months
  The improvement in The American Orthopaedic Foot & Ankle Society (AOFAS) score from the baseline was observed at 12 months after injury on a scale of 0-100.

SECONDARY OUTCOMES:
Signs of healing on X-ray at 6 weeks | 6 weeks
  The presence or absence of signs of healing on X-ray were observed at 6 weeks after injury.
Signs of healing on X-ray at 12 months | 6 weeks
  The presence or absence of signs of healing on X-ray were observed at 12 months after injury.
Extremity loading | 6 weeks
  The ability to load the injured extremity was measured in per cent of full loading.

CONTACTS AND LOCATIONS:
Overall Officials: Jiří Demel, MD, Principal Investigator — University Hospital Ostrava; Leopold Pleva, Ass.Prof.,MD,CSc., Study Director — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
The researchers do not plan to share individual participant data with other researchers.

REFERENCES:
- [Background] Dameron TB Jr. Fractures and anatomical variations of the proximal portion of the fifth metatarsal. J Bone Joint Surg Am. 1975 Sep;57(6):788-92. PMID 1099103
- [Background] Kavanaugh JH, Brower TD, Mann RV. The Jones fracture revisited. J Bone Joint Surg Am. 1978 Sep;60(6):776-82. PMID 701310
- [Background] Landorf KB. Clarifying proximal diaphyseal fifth metatarsal fractures. The acute fracture versus the stress fracture. J Am Podiatr Med Assoc. 1999 Aug;89(8):398-404. doi: 10.7547/87507315-89-8-398. PMID 10466292
- [Background] Malkus T, Soukup B. [Jones fracture.]. Acta Chir Orthop Traumatol Cech. 1999;66(1):15-21. Czech. PMID 20478127
- [Background] Marshall PD, Evans PD, Richards J. Laboratory comparison of the cannulated Herbert bone screw with ASIF cancellous lag screws. J Bone Joint Surg Br. 1993 Jan;75(1):89-92. doi: 10.1302/0301-620X.75B1.8421045.
- [Background] Mindrebo N, Shelbourne KD, Van Meter CD, Rettig AC. Outpatient percutaneous screw fixation of the acute Jones fracture. Am J Sports Med. 1993 Sep-Oct;21(5):720-3. doi: 10.1177/036354659302100514. PMID 8238714
- [Background] Nunley JA. Fractures of the base of the fifth metatarsal: the Jones fracture. Orthop Clin North Am. 2001 Jan;32(1):171-80. doi: 10.1016/s0030-5898(05)70200-5. PMID 11465126
- [Background] Pietropaoli MP, Wnorowski DC, Werner FW, Fortino MD. Intramedullary screw fixation of Jones fractures: a biomechanical study. Foot Ankle Int. 1999 Sep;20(9):560-3. doi: 10.1177/107110079902000904. PMID 10509682
- [Background] Quill GE Jr. Fractures of the proximal fifth metatarsal. Orthop Clin North Am. 1995 Apr;26(2):353-61. PMID 7724197
- [Background] Rosenberg GA, Sferra JJ. Treatment strategies for acute fractures and nonunions of the proximal fifth metatarsal. J Am Acad Orthop Surg. 2000 Sep-Oct;8(5):332-8. doi: 10.5435/00124635-200009000-00007. PMID 11029561
- [Background] STEWART IM. Jones's fracture: fracture of base of fifth metatarsal. Clin Orthop. 1960;16:190-8. No abstract available. PMID 13834594